CLINICAL TRIAL: NCT06085586
Title: Evaluation of Safety and Performance Outcomes of the Fibulink Syndesmosis Repair System With Early Full-Weight Bearing
Brief Title: Fibulink Syndesmosis Repair System With Early Full-Weight Bearing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-08-15-MMC
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Ankle Fractures; Bimalleolar Fractures; Syndesmotic Injuries; Bimalleolar Equivalent Fracture; Maisonneuve Fracture; Trimalleolar Fractures; Ankle Dislocation
Keywords: Ankle Fractures; Bimalleolar Fractures; Bimalleolar Equivalent Fracture; Trimalleolar Fractures; Maisonneuve Fractures; Syndesmotic Injuries; Ankle Dislocations
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries; Fibula Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1) Early Full Weight Bearing (Experimental): Full weight bearing (100%) initiated at 4 weeks postoperatively
  Interventions: Other: Early Weight Bearing
- 2) Normal Full Weight Bearing (Active Comparator): Full weight bearing (100%) initiated at 6 weeks postoperatively
  Interventions: Other: Normal Weight Bearing

INTERVENTIONS:
Other: Early Weight Bearing — Full weight bearing (100%) initiated at 4 weeks postoperatively
  Arms: 1) Early Full Weight Bearing
Other: Normal Weight Bearing — Full weight bearing (100%) initiated at 6 weeks postoperatively
  Arms: 2) Normal Full Weight Bearing

SUMMARY:
The purpose of the study is to evaluate the ability of the Fibulink Syndesmosis Repair System to maintain reduction of the ankle syndesmosis. Appropriate reduction of the syndesmosis is critical due the changes in tibiotalar contact pressure observed in cadaveric studies.6,7 Malreduction and instability of the distal tibiotalar joint can lead to chronic instability, increased articular damage and ultimately degenerative arthritis.7,8 Medial to lateral translation of distal tibia and fibula of 2 mm or more has been considered pathologic.9 Earlier biomechanical study demonstrated the Fibulink system is superior in maintaining displacement of less than 2 mm.4 Given the improved strength, we also look to evaluate the outcomes of initiating full weight bearing (100%) with Controlled Ankle Motion (CAM) boot at 4 weeks postoperatively. One of the big limitations for trans-osseous screw fixation is delayed weight bearing due to risk of screw breakage.1 Suture button technique allowed for early weight bearing with average of 6 weeks postoperatively using TightRope.2,10-12By initiating full weight bearing (100%) with CAM boot at 4 weeks postoperatively, this would be a significant improvement in current clinical practice.

DETAILED DESCRIPTION:
All ankle fractures will be evaluated by the orthopedic team. Standard radiographs including anteroposterior (AP), lateral and mortise view of the ankle will be obtained. Manual or gravity stress view will be performed if needed. Treatment options including nonoperative and operative management will be discussed with the patient including the risks and benefits. An informed decision will be made. Two separate informed consent will be obtained. The first will be an informed consent for the surgery, detailing the planned surgical procedure. The second will be an informed consent for the enrollment of the study, detailing the purpose of the study and the use of the Fibulink Syndesmotic Repair System in any cases of syndesmotic injury.

Should the patient elects to proceed with surgery, the patient will be informed that fixation of the fractures will be performed first. Direct lateral approach to the distal fibular will be used for fixation of the lateral malleolus. If necessary, direct medial approach will be used for fixation of the medial malleolus. Once the fractures have been fixed, the syndesmosis will be stressed intraoperatively under live fluoroscopy. Based on the parameters described in 6.3, a decision will be made whether fixation of the syndesmosis is required if instability is noted. If fixation of the syndesmosis is required, it will be performed through the direct lateral approach.

The research coordinator will be informed of all patients that had the syndesmosis fixed with the Fibulink System. Patients will then be followed at the following time points: 2 weeks, 4-6 weeks, 8-10 weeks, 3 months and 6 months. During each follow-up time points, the tibiofibular overlap, tibiofibular clear space and medial clear space will be measured and recorded. The postoperative protocol will be as follow: Immediately post-op, patient will be placed in a short leg cast. At 2 weeks postop, the short leg cast will be removed. Suture removal will be performed. Patient will be placed in a CAM boot and instructed to perform early active ankle range-of-motion. Depending on the study group, at 4 weeks or 6 weeks postop, full weight bearing (100%) in the CAM boot will be allowed. Physical therapy will begin. At 8-10 weeks postop, full weight bearing (100%) without CAM boot will begin. Patients will continue to follow-up at 3 months and 6 months.

The research coordinator will ensure proper follow-up and will be responsible for data collection and input. After achieving the planned number of participants, the results of the two study sites will be gathered. Appropriate statistical analysis will be performed, and the results will be presented in a full manuscript format.

ELIGIBILITY:
Inclusion Criteria:

* ankle fracture with syndesmotic disruption as assessed with intra-operative cotton test.

This includes the following injuries:

* Syndesmotic sprain (without fractures)
* Bimalleolar equivalent ankle fractures
* Bimalleolar ankle fractures
* Maisonneuve fractures
* Trimalleolar ankle fractures without the need for posterior malleolus fixation
* Ankle fracture dislocations

Exclusion Criteria:

* 1) previous ankle surgery, 2) active local infection about the ankle, 3) chronic ankle deformity secondary to trauma or congenital, 4) ligamentous laxity, 5) pathologic fractures, 6) peripheral vascular disease, 7) peripheral neuropathy, 8) diabetes neuropathy and charcot, 9) open fractures, 10) poly trauma, 11) inability to provide informed consent, 12) symptomatic ankle osteoarthritis, 12) retained hardware, 13) pregnant, 14) metabolic bone disease, 15) history of chronic steroid use, 16) mal-reduced ankle fractures

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
6 Month Reduction Quality | 6 Months
  The primary objective is to evaluate the reduction and maintenance of the reduction of ankle syndesmosis in 6 months after initiating full weight bearing (100%) at 4 weeks or 6 weeks postoperatively. This will be determined based on comparing the tibiofibular overlap, tibiofibular clear space and medial clear space preoperative values.

SECONDARY OUTCOMES:
2 Week Reduction Quality | 2 Weeks
  Reduction and maintenance of the reduction of the ankle syndesmosis at 2 weeks based on the tibiofibular overlap, tibiofibular clear space and medial clear space preop values.
4-6 Week Reduction Quality | 4-6 Weeks
  Reduction and maintenance of the reduction of the ankle syndesmosis at 4-6 weeks based on the tibiofibular overlap, tibiofibular clear space and medial clear space preop values.
8-10 Week Reduction Quality | 8-10 Weeks
  Reduction and maintenance of the reduction of the ankle syndesmosis at 8-10 weeks based on the tibiofibular overlap, tibiofibular clear space and medial clear space preop values.
3 Month Reduction Quality | 3 Months
  Reduction and maintenance of the reduction of the ankle syndesmosis at 3 months based on the tibiofibular overlap, tibiofibular clear space and medial clear space preop values.
Reoperation or Revision | 6 Months
  Unplanned Reoperation or late-stage revision
OR Time | 1 Day
  Operating Room Time in Minutes
Surgical Approach/Procedure Type | 1 Day
  Surgical Approach/Procedure Type
Type of Additional Fixation | 1 Day
  Type of Additional Fixation
Intraoperative Complications | 1 Day
  Any complications that occurred intraoperatively
Postoperative Complications | 30 Days
  Any complications that occurred postoperatively within 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Abdelgawad, MD PhD MBA, Principal Investigator — Vice Chair of Orthopedic Clinical Programs, Director of Pediatric Orthopedic Surgery
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thornes B, Shannon F, Guiney AM, Hession P, Masterson E. Suture-button syndesmosis fixation: accelerated rehabilitation and improved outcomes. Clin Orthop Relat Res. 2005 Feb;(431):207-12. PMID 15685077
- [Background] Degroot H, Al-Omari AA, El Ghazaly SA. Outcomes of suture button repair of the distal tibiofibular syndesmosis. Foot Ankle Int. 2011 Mar;32(3):250-6. doi: 10.3113/FAI.2011.0250. PMID 21477543
- [Background] Morellato J, Louati H, Bodrogi A, Stewart A, Papp S, Liew A, Gofton W. The Effect of Varying Tension of a Suture Button Construct in Fixation of the Tibiofibular Syndesmosis-Evaluation Using Stress Computed Tomography. J Orthop Trauma. 2017 Feb;31(2):103-110. doi: 10.1097/BOT.0000000000000737. PMID 28129269
- [Background] Dynamic and Load-to-Failure Testing of the DePuy Synthes FIBULINK TM Syndesmosis Repair System and Arthrex Syndesmosis TightRope ® XP Implant System Materials and Methods. 2020.
- [Background] Desai S. Syndesmosis Repair: 14 Patient Case Series.
- [Background] Ramsey PL, Hamilton W. Changes in tibiotalar area of contact caused by lateral talar shift. J Bone Joint Surg Am. 1976 Apr;58(3):356-7. PMID 1262367
- [Background] Hunt KJ, Goeb Y, Behn AW, Criswell B, Chou L. Ankle Joint Contact Loads and Displacement With Progressive Syndesmotic Injury. Foot Ankle Int. 2015 Sep;36(9):1095-103. doi: 10.1177/1071100715583456. Epub 2015 May 6. PMID 25948693
- [Background] Porter DA, Jaggers RR, Barnes AF, Rund AM. Optimal management of ankle syndesmosis injuries. Open Access J Sports Med. 2014 Aug 5;5:173-82. doi: 10.2147/OAJSM.S41564. eCollection 2014. PMID 25177153
- [Background] Hunt KJ. Syndesmosis injuries. Curr Rev Musculoskelet Med. 2013 Dec;6(4):304-12. doi: 10.1007/s12178-013-9184-9. PMID 23949902
- [Background] Cottom JM, Hyer CF, Philbin TM, Berlet GC. Transosseous fixation of the distal tibiofibular syndesmosis: comparison of an interosseous suture and endobutton to traditional screw fixation in 50 cases. J Foot Ankle Surg. 2009 Nov-Dec;48(6):620-30. doi: 10.1053/j.jfas.2009.07.013. Epub 2009 Sep 15. PMID 19857816
- [Background] Thornes, Brian FRCSI; McCartan, Damien MB. Ankle Syndesmosis Injuries Treated with the TightRopeTM Suture-Button Kit. Techniques in Foot & Ankle Surgery 5(1):p 45-53, March 2006.
- [Background] Latham AJ, Goodwin PC, Stirling B, Budgen A. Ankle syndesmosis repair and rehabilitation in professional rugby league players: a case series report. BMJ Open Sport Exerc Med. 2017 Apr 1;3(1):e000175. doi: 10.1136/bmjsem-2016-000175. eCollection 2017. PMID 28761696
- [Background] Cotton FJ. Dislocations and Joint-Fractures. Philadelphia: W. B. Saunders Company, 1910.
- [Background] Ebraheim NA, Lu J, Yang H, Mekhail AO, Yeasting RA. Radiographic and CT evaluation of tibiofibular syndesmotic diastasis: a cadaver study. Foot Ankle Int. 1997 Nov;18(11):693-8. doi: 10.1177/107110079701801103. PMID 9391813
- [Background] Harper MC, Keller TS. A radiographic evaluation of the tibiofibular syndesmosis. Foot Ankle. 1989 Dec;10(3):156-60. doi: 10.1177/107110078901000308. PMID 2613128
- [Background] Leeds HC, Ehrlich MG. Instability of the distal tibiofibular syndesmosis after bimalleolar and trimalleolar ankle fractures. J Bone Joint Surg Am. 1984 Apr;66(4):490-503. PMID 6423645
- [Background] Rigby RB, Cottom JM. Does the Arthrex TightRope(R) provide maintenance of the distal tibiofibular syndesmosis? A 2-year follow-up of 64 TightRopes(R) in 37 patients. J Foot Ankle Surg. 2013 Sep-Oct;52(5):563-7. doi: 10.1053/j.jfas.2013.04.013. Epub 2013 Jun 14. PMID 23770192
- [Background] Mukhopadhyay S, Metcalfe A, Guha AR, Mohanty K, Hemmadi S, Lyons K, O'Doherty D. Malreduction of syndesmosis--are we considering the anatomical variation? Injury. 2011 Oct;42(10):1073-6. doi: 10.1016/j.injury.2011.03.019. Epub 2011 May 6. PMID 21550047

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT06085586/Prot_SAP_000.pdf